CLINICAL TRIAL: NCT04960644
Title: A Multi-cohort, Phase Ⅲ Study of Methotrexate Combined Corticosteroid as First-line Therapy in Chinese Patients With Acute Graft vs. Host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: MTX and Steroid as First-line Therapy for aGVHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Chief of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-202105-K3-01
Record Dates: First submitted 2021-06-23; First posted 2021-07-14 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Acute GVH Disease
Keywords: acute GVHD; MTX; Corticosteroid
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MTX and corticosteroid (Experimental): perimental: MTX and corticosteroid Methylprednisolone 1 mg/kg/day was given for 10 days and then gradually reduce the dose according to patient's response MTX (5-6mg/m^2/day,Maximum dose 10mg/day) was given on days 1, 3, and 8, and repeated weekly until aGVHD was CR
  Interventions: Drug: MTX
- corticosteroid (Active Comparator): perimental: corticosteroid Methylprednisolone 1 mg/kg/day was given for 10 days and then gradually reduce the dose according to patient's response
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: MTX — MTX (5-10 mg/day,Dmax 10mg/day) was given on days 1, 3, and 8, and repeated weekly until aGVHD was CR
  Other Names: Corticosteroid
  Arms: MTX and corticosteroid
Drug: Corticosteroid — corticosteroid Methylprednisolone 1 mg/kg/day was given for 10 days and then the dosage was gradually reduced according to patient's response
  Arms: corticosteroid

SUMMARY:
The aim of the study is to identify the efficacy and safety of methotrexate (MTX) combined corticosteroid as first-line therapy for acute graft-versus-host disease (aGVHD) after allogeneic hematopoietic stem cell transplantation (alloHSCT).

DETAILED DESCRIPTION:
Allo-HSCT is an effective treatment of malignant hematopoietic diseases. However, aGVHD remains a major complication after allo-HSCT and the destruction of recipient tissues by alloantigen-activated T cells is a key event in the development of aGVHD. Corticosteroid is the standard first-line therapy for aGVHD due to their roles in suppressing T cell responses. However, the response rate of corticosteroid was approximate 50%, and the clinical outcomes of patients with corticosteroid refractory GVHD were poor. Thus far, no combination therapy had been prove to be superior to corticosteroid alone as initial therapy for aGVHD. The study hypothesis: MTX combined corticosteroid treatment could help to further ameliorate the activity of T cells and control aGVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are fully informed and sign informed consent by themselves or their guardians;
2. Patients receiving allogeneic hematopoietic stem cell transplantation;
3. Patients with acute graft-versus-host disease of grade II-IV were diagnosed after transplantation;
4. Patients with stable implantation of granulocytes and platelets.
5. ECOG score ≤3

Exclusion Criteria:

1. Patients with severe brain, heart, kidney or liver dysfunction unrelated to graft-versus host disease;
2. Patients with uncontrollable active infection;
3. Patients with recurrence of primary malignant hematopathy;
4. Expected survival is less than 3 months
5. Patients who have histories of severe allergic reactions
6. Pregnant or lactating women
7. The researcher judges that there are other factors that are not suitable for participating

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) for aGVHD treatment after treatment | 10 days
  Overall response rate is defined as the proportion of patients demonstrating a complete response or partial response without requirement for additional systemic therapies for an earlier progression, mixed response or non-response

SECONDARY OUTCOMES:
Overall response rate (ORR) for aGVHD treatment at 28 days after treatment | 28 days
  Overall response rate is defined as the proportion of patients demonstrating a complete response or partial response without requirement for additional systemic therapies for an earlier progression, mixed response or non-response
Overall response rate (ORR) for aGVHD treatment at 42 days after treatment | 42 days
  Overall response rate is defined as the proportion of patients demonstrating a complete response or partial response without requirement for additional systemic therapies for an earlier progression, mixed response or non-response
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 42 days
  Data collection including questionnaires at individual and group visits and physician interviews at individual visits will be used to assess participants for treatment-related adverse events.
cGVHD | 1 years
  The cumulative incidence of chronic GVHD
Infection and poor graft function | 1 year
  The cumulative incidence of severe infection and poor graft function
Relapse | 1 year
  The cumulative incidence of relapse
Non-relapse mortality | 1 year
  The cumulative incidence of non-relapse mortality
Overall survival | 1 year
  The cumulative incidence of overall survival
Disease free survival | 1 year
  The cumulative incidence of disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, Dr., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Liu QF, Wu DP, Xu ZL, Han TT, Sun YQ, Huang F, Fan ZP, Xu N, Chen F, Zhao Y, Kong Y, Mo XD, Xu LP, Zhang XH, Liu KY, Huang XJ. Mini-dose methotrexate combined with methylprednisolone for the initial treatment of acute GVHD: a multicentre, randomized trial. BMC Med. 2024 Apr 25;22(1):176. doi: 10.1186/s12916-024-03395-y. PMID 38664766